CLINICAL TRIAL: NCT07365267
Title: Study on the Cosmetic Outcome and Safety Evaluation of 3D Printed Biodegradable Biological Mesh for One-Stage Breast Reconstruction After Radical Mastectomy :A Prospective, Single-Center, Single-Arm Clinical Study
Brief Title: Study on the Cosmetic Outcome and Safety Evaluation of 3D Printed Biodegradable Biological Mesh for One-Stage Breast Reconstruction After Radical Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Zhang Juliang-1, Associate Chief Physician, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20252568-F-1
Record Dates: First submitted 2026-01-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Breast Reconstruction After Mastectomy; 3D-Printed Biodegradable Biological Mesh
Keywords: 3D-Printed Biodegradable Biological Mesh; breast reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D printing patient (Experimental): immediate breast reconstruction using 3D-Printed Biodegradable Biological Mesh combined with a silicone breast prosthesis
  Interventions: Procedure: Implantation of a silicone breast prosthesis combined with a 3D-printed biodegradable mesh

INTERVENTIONS:
Procedure: Implantation of a silicone breast prosthesis combined with a 3D-printed biodegradable mesh — Nipple-sparing subcutaneous mastectomy combined with an implant for immediate breast reconstruction will be performed according to standard clinical practice. The choice of incision will be at the surgeon's discretion. Intraoperatively, tissue from behind the nipple will be sent for frozen section histopathological examination. If the margin is positive, the nipple-areolar complex will be resected following safety principles. The 3D-printed biodegradable biological mesh will be used to wrap the silicone implant, which is then placed in the subcutaneous tissue. The wound will be soaked and irrigated with sterile distilled water and normal saline. After achieving thorough hemostasis, a drain will be placed, and the skin will be closed in layers.

SUMMARY:
Primary objective of this trial: To evaluate the clinical performance (aesthetic outcome and quality of life) and safety of a 3D-printed biodegradable biological mesh in post-mastectomy immediate breast reconstruction. The study targets adult women undergoing total mastectomy for breast cancer followed by implant-based reconstruction. It aims to determine the utility of the 3D-printed biodegradable mesh in implant-based breast reconstruction, assess its influence on tissue regeneration, postoperative cosmetic result, and complication profile.

DETAILED DESCRIPTION:
Study Objectives

* Primary Objective: To evaluate the clinical efficacy and safety of breast reconstruction using a 3D- printed biodegradable biological mesh.
* Secondary Objective: To evaluate the postoperative quality of life and breast cancer-free interval after breast reconstruction with a 3D-printed biodegradable biological mesh.

Treatment Plan

* Study Enrollment and Informed Consent: All subjects will sign the relevant informed consent forms before surgery.
* Preoperative Assessment: Patients will complete the Chinese version of the BREAST-Q V2.0 scale and the QoL (Quality of Life) scale.
* Preoperative Imaging Assessment:

Enrolled patients will undergo a preoperative thin-slice breast MRI (3.0T) using a multi-channel phased-array dedicated breast coil. The patient will be in a prone position, head-first. The operator will assist in placing the breast in the center of the coil, allowing it to hang naturally without compression to maintain its natural shape. The prone position also helps reduce respiratory motion artifacts. The patient's arms will be placed naturally in front of their head, avoiding the scan field to reduce artifacts. A high-pressure injector will be connected to an intravenous catheter. An axial three-dimensional thin- slice scan will be selected to display both breasts simultaneously, showing the radially arranged ducts converging towards the nipple and the glandular tissue in the axillary tail. The 3D thin-slice scan facilitates sagittal and coronal reconstructions. The scan range will cover the superior and inferior borders of both breasts.

Conventional Plain Scan: A SE T1WI sequence will be used to obtain T1-weighted transverse images. Scan parameters: TR 500ms, TE 15ms, slice thickness 2.8mm, FOV for both breasts 360mm, matrix 256x320, NEX 2.

Functional Imaging: A FLASH (Fast Low Angle Shot) sequence will be used for 3D dynamic contrast-enhanced scanning. Scan parameters: TR 4.42ms, TE 1.41ms, flip angle 12 degrees, FOV for both breasts 360mm, matrix 512x384, slice thickness 1.2mm, 6 acquisitions, total time 6 minutes 19 seconds, one acquisition 55 seconds. The contrast agent will be Gd-DTPA at a dose of 0.2 mmol/kg, administered as a bolus injection via an antecubital or dorsal hand vein at a rate of 3 ml/s, followed by a 20 ml saline flush at the same rate. After the first scan, the automatic high-pressure injector will be activated to inject the Gd-DTPA contrast agent and saline. The enhanced scan will be initiated simultaneously with the injection and repeated 5 times. The post-enhancement images will be subtracted from the initial plain scan images to obtain 5 sets of subtracted images. These subtracted images will then be reconstructed using the Maximum Intensity Projection (MIP) method to generate 5 three-dimensional enhanced images.

* Preoperative Implant Size Assessment: The implant volume will be estimated using empirical methods to determine the proposed implant size.
* Surgical Simulation, Design, and 3D Printing of PCL Mesh:

Using medical-grade polycaprolactone (PCL) microspheres as the printing material, the optimized breast mesh model will be manufactured using Selective Laser Sintering (SLS) technology. The model data will be processed by slicing software, and the processed data will be input into the SLS printer. The SLS printer will control the laser scanning path according to the contour and filling structure of the current layer to sinter the PCL powder. This process is repeated layer by layer to print the model structure. After printing, the structure is removed, residual powder on the surface is cleaned off, and the final product is sterilized with low-temperature ethylene oxide for 48 hours before use.

* Surgery:Nipple-sparing subcutaneous mastectomy combined with an implant for immediate breastreconstruction will be performed according to standard clinical practice. The choice of incision will be at the surgeon's discretion. Intraoperatively, tissue from behind the nipple will be sent for frozen section histopathological examination. If the margin is positive, the nipple-areolar complex will be resected following safety principles. The 3D-printed biodegradable biological mesh will be used to wrap the silicone implant, which is then placed in the subcutaneous tissue. The wound will be soaked and irrigated with sterile distilled water and normal saline. After achieving thorough hemostasis, a drain will be placed, and the skin will be closed in layers.
* Postoperative Management:Electronic health records will be established. Follow-ups will be conducted at 1 week, 1 month, 3 months, 6 months, and 12 months post-surgery, and then every 6 months thereafter. Follow-up content includes recording complications or adverse reactions, completing the Chinese version of the BREAST-Q V2.0 scale for breast aesthetics, satisfaction, and QoL assessment, and monitoring for metastasis or recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients aged 18 to 70 years.
* Histopathologically confirmed invasive breast cancer, as defined by the latest ASCO/NCCN guidelines.
* Unable to undergo breast-conserving surgery or willing to undergo total mastectomy with immediate implant-based breast reconstruction.
* ECOG performance status of 0-1.
* Voluntary participation in the study and signing of the written informed consent form.

Exclusion Criteria:

* Age >70 years.
* Metastatic breast cancer (Stage IV) at initial diagnosis.
* Multicentric, extensive, diffuse lesions, or inflammatory breast cancer.
* Tumor involvement of the nipple-areolar complex.
* Breast cancer during pregnancy.
* History of other malignancies within the past 5 years, except for cured cervical carcinoma in situ or non-melanoma skin cancer.
* Abnormal function of vital organs such as heart, lungs, liver, or kidneys; poorly controlled diabetes, etc., rendering the patient unable to tolerate surgery.
* Patients deemed unsuitable for participation by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
postoperative cosmetic results and safety | At 1 week, 1 month, 3 months, 6 months, 12 months ，18 months，and 24 months post-surgery，through study completion, an average of 2 year.
  Postoperative Cosmetic Outcome and Safety: Patient satisfaction will be scored using the reconstruction module of the Breast-Q questionnaire, which includes satisfaction with breasts, satisfaction with surgical outcome, and satisfaction with treatment. Satisfaction with breasts will be the primary endpoint of this study. After the BREAST-Q questionnaire is completed, its score, known as the Q-SCORE, will be calculated. The specific evaluation requires the use of Q-SCORE scoring software. The Breast-Q scale also includes scores for satisfaction with surgery, satisfaction with treatment, and health-related quality of life (QOL), covering physical, psychosocial, and sexual well-being. For all dimensions, a higher patient-reported score indicates higher satisfaction and better quality of life.In outcome of BREAST-Q questionnaire, BREAST-Q scales (domains) are scored on a 0-100 range, with higher scores indicating greater satisfaction or better health-related quality of life.

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | At 1 week, 1 month, 3 months, 6 months, 12 months ，18 months，and 24 months post-surgery，through study completion, an average of 2 year.
  Recurrence in the ipsilateral breast, chest wall, skin, or surgical scar confirmed by imaging is defined as "local recurrence day" on the date of the earliest imaging finding. If local recurrence is diagnosed based on clinical history and physical examination, the date of clinical determination is the "local recurrence day." If diagnosed by cytology or histopathology, the date of the earliest examination is the "local recurrence day." RFS is the time from the date of surgery to the date of disease recurrence or death. For patients with no observed recurrence or death, the follow-up is censored at the date of the last confirmation of no recurrence. An increase in tumor markers such as CEA alone is not sufficient to diagnose recurrence.
Disease-Free Survival (DFS) | At 1 week, 1 month, 3 months, 6 months, 12 months ，18 months，and 24 months post-surgery，through study completion, an average of 2 year.
  The time from the date of surgery to the date of tumor recurrence (if the specific date of recurrence is unknown, the date of death due to the tumor is used). For patients with no observed recurrence or death, the follow-up is censored at the date of the last confirmation of no recurrence (last date of no recurrence confirmation: the last date of outpatient visit or examination).
Overall Survival (OS) | At 1 week, 1 month, 3 months, 6 months, 12 months ，18 months，and 24 months post-surgery，through study completion, an average of 2 year.
  The time from the date of surgery to death from any cause (if death has not occurred, the time to the last follow-up). For surviving patients, the follow-up is censored at the date of the last confirmation of survival. For patients lost to follow-up, it is censored at the last date of confirmed survival before being lost.
Surgical Technical Safety (Complication Rate) | At 1 week, 1 month, 3 months, 6 months, 12 months ，18 months，and 24 months post-surgery，through study completion, an average of 2 year.
  Intraoperative complications: Including but not limited to: intraoperative bleeding, major vessel injury, subcutaneous emphysema, hypercapnia, etc. The rate is calculated as the number of patients with any intraoperative complication divided by the total number of patients who underwent surgery.
  Postoperative complications: Including but not limited to: infection, skin flap or nipple-areolar complex necrosis, sensory abnormalities in the surgical area, mesh-related complications, etc. The rate is calculated as the number of patients with any postoperative complication divided by the total number of patients who underwent surgery.
  Unplanned reoperation rate: The proportion calculated as the number of patients undergoing unplanned reoperation divided by the total number of patients who underwent surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of the Air Force Medical University, Xi'an, Shaanxi, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: in English (2025-12-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT07365267/Prot_SAP_000.pdf
  • Informed Consent Form: in English (2025-12-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT07365267/ICF_001.pdf